CLINICAL TRIAL: NCT00002435
Title: Study of the Activity of Thymic Humoral Factor (THF Gamma 2) on HIV Load in HIV-Positive Individuals With CD4+ Cell Counts in the Range of 200-500 Cells/mm3
Brief Title: A Study of Thymic Humoral Factor (THF Gamma 2) in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacia (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 136A; CS 112010-999
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-02

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Antiviral Agents; Zidovudine; thymic humoral factor gamma 2
MeSH Terms: conditions — HIV Infections | interventions — thymic humoral factor; Zidovudine

INTERVENTIONS:
Drug: Thymic Humoral Factor
Drug: Zidovudine

SUMMARY:
To investigate the safety of thymic humoral factor (THF gamma 2), its effect on HIV load based on at least a 75 percent decrease in HIV quantitative PCR RNA copies/ml, and its persistence when administered in combination with an antiretroviral nucleoside derivative (zidovudine; AZT). To assess the effects of THF gamma 2 on T-cells, quality of life, and progression of disease.

DETAILED DESCRIPTION:
All patients receive 12 weeks of AZT before being randomized to self-administer one of two doses of THF gamma 2 or placebo for 15 consecutive days and then twice weekly for an additional 50 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* AZT or another antiretroviral agent (marketed or investigational under a Treatment IND).
* Primary prophylaxis for Pneumocystis carinii pneumonia (PCP), toxoplasmosis, and Mycobacterium avium-intracellulare (MAI) if patient's CD4 count decreases to < 200 cells/mm3.
* Other marketed drugs as required.

Patients must have:

* HIV seropositivity and be either asymptomatic or have persistent generalized lymphadenopathy (PGL).
* No history of symptoms in Category B or C of 1993 Case Definition, other than oral candidiasis following previous broad-spectrum antibiotic therapy.
* Mean CD4 of 200-500 cells/mm3.
* HIV-1 positive PCR RNA.
* Ability to self-administer study drug by IM injection.
* Ability to tolerate AZT at 600 mg daily during first 8 weeks of run-in period (if AZT naive) OR tolerated AZT at >= 500 mg daily for at least 3 months but no more than 12 months prior to randomization.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malignancy.
* Hematuria.
* Proteinuria > 1+.

Concurrent Medication:

Excluded:

* Non-antiretroviral agents with known or suspected activity against HIV.
* Investigational new drugs that are not antiretroviral agents distributed under a Treatment IND.

Patients with the following prior conditions are excluded:

Myositis within the past 6 months.

Prior Medication:

Excluded:

* Experimental therapy, including interleukin-2, interferon, erythropoietin, or filgrastim nucleoside within 6 weeks prior to study entry.
* Prior antiretroviral therapy (AZT-naive patients only).

Prior Treatment:

Excluded within 6 weeks prior to study entry:

* Blood transfusion or blood products. Active alcoholism, drug abuse, or a mental or psychiatric problem sufficient to prevent adequate compliance with study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - UCI, Irvine, California
  - Southwest Community Based AIDS Treatment Group - COMBAT, Los Angeles, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - Gottlieb Med Group, Sherman Oaks, California
  - Mem Hosp Hollywood, Hollywood, Florida
  - Goodgame Med Group, Maitland, Florida
  - Chelsea Village Med Ctr, New York, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Dr Alfred F Burnside Jr, Columbia, South Carolina
  - Infectious Disease Physicians Inc, Annandale, Virginia